CLINICAL TRIAL: NCT06032741
Title: Prognosis in Patients With Guillain-Barre Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GBS
Record Dates: First submitted 2022-12-26; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-12

CONDITIONS: Guillain-Barre Syndrome
Keywords: Guillain-Barre Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mechanical ventilation group: Patients with Guillain-Barré Syndrome require mechanical ventilation during hospitalization
- no mechanical ventilation group: Patients with Guillain-Barré Syndrome do not require mechanical ventilation during hospitalization

SUMMARY:
The goal of this observational study is to explore significant indicators to predict the early prognosis and late prognosis in patients with Guillain-Barre syndrome.

DETAILED DESCRIPTION:
This is a multicenter study(approximately three) with over 450 subjects.Clinical data were collected by consulting the patient's electronic history. The data included demographic information, blood biochemical markers, clinical characteristics and electromyography. All participants provided their written informed consent to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilled clinical, biological, and electrophysiology criteria for Guillain-barre syndrome.

Exclusion Criteria:

* nonidiopathic Guillain-barre syndrome and Miller Fisher syndrome

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a multicenter study(approximately three) with over 450 subjects.Clinical data were collected by consulting the patient's electronic history. The data included demographic information, blood biochemical markers, clinical characteristics and electromyography. All participants provided their written informed consent to participate in this study.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2013-01-02 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
the severity of Guillain-barre syndrome | baseline, at 1 week, at 26 weeks
  The Guillain-Barre syndrome disability score is a wide scale for the severity of Guillain-Barre syndrome (0, optimal health; 1, minor symptoms, able to run; 2, able to walk unaided 10 m, unable to run; 3, able to walk 10 m across an open space with help; 4 bedridden or wheelchair users; 5, require assisted ventilation; 6, dead)(deceased).The higher the score, the worse the prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China